CLINICAL TRIAL: NCT00270283
Title: A Double-Blind, Placebo-Controlled Study With Open-Label Follow-up to Determine the Safety and Efficacy of Subcutaneous Doses of r-HuEPO in AIDS Patients With Anemia Induced by Their Disease and AZT Therapy
Brief Title: A Study to Evaluate the Safety and Efficacy of Epoetin Alfa Versus Placebo for the Treatment of Anemia in Patients With Acquired Immunodeficiency Syndrome (AIDS) Who Are Receiving Zidovudine (AZT) Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006076; NCT00473759 (obsolete NCT alias)
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2009-07

CONDITIONS: Acquired Immunodeficiency Syndrome; Anemia
Keywords: Anemia; AIDS; erythropoietin; epoetin alfa; Quality of Life; Zidovudine; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of epoetin alfa in AIDS patients for the treatment of anemia that is a result of the disease and zidovudine (AZT) treatment. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
It is estimated that approximately 75% to 80% of patients with AIDS experience anemia, which can be caused by AIDS or by the therapy patients receive for AIDS treatment (for example, zidovudine [AZT]). Anemia is a condition in which a patient has below normal levels of hemoglobin, the substance in red blood cells that carries oxygen to all parts of the body. People with severe anemia may experience fatigue and shortness of breath with activity. Therefore, this condition can have a negative influence on a person's quality of life. Epoetin alfa, used to treat anemia, is a genetically engineered form of a natural hormone, erythropoietin, that stimulates red blood cell production. This is a randomized, double-blind, placebo-controlled, parallel group study with an open-label follow-up period that is designed to evaluate the safety and effectiveness of epoetin alfa treatment in patients with AIDS who are being treated with AZT. The study consists of 3 periods: a screening period to determine if patients are eligible for the study, a double-blind treatment period, and an open-label treatment period. Eligible patients will be randomly assigned to one of two groups: epoetin alfa 150 units per kilogram or matching placebo. Patients will be treated with study medication (injected under the skin) 3 times a week for 12 weeks, or until their hematocrit reaches 38% to 40%. In the open-label period, all patients receive epoetin alfa injected under the skin for up to 6 months. Effectiveness will be determined by the change in hemoglobin and hematocrit (laboratory tests used to evaluate the severity of anemia), transfusion requirements, the patient's quality of life assessment, and the physician's global evaluation of the drug effect. Safety assessments include the incidence and severity of adverse events during the study, changes in clinical laboratory tests (hematology, biochemistry, and urinalysis), vital signs, electrocardiograms (ECGs), and physical examination findings. The study hypothesis is that AIDS patients who are receiving AZT and who are treated with epoetin alfa will have a lower incident of anemia compared with patients receiving placebo.

Double-blind: epoetin alfa, 150 units per kilogram [U/kg] of body weight, or placebo, injected under the patient's skin 3 times a week for 12 weeks or until the hematocrit level reaches 38% to 40%. Open-label: epoetin alfa, 200 U/kg, 3 times a week for up to 6 months (once weekly after hematocrit reaches 38% to 40%). Dose may be adjusted up to 1500 U/kg per week, as needed.

ELIGIBILITY:
Inclusion Criteria: - Patients with a confirmed diagnosis of AIDS - having a Performance score of 0, 1, or 2 (patients' ability to perform daily activities, a score ranging from 0 [fully active, no disease restriction] to 3 [capable of only limited self-care, confined to bed or chair more than 50% of waking hours]) - taking a maintenance dose of AZT of at least 400 mg/day - having a hematocrit of at least 30% and a history of a >=15% decrease in hematocrit since starting AZT therapy, or have become dependent on transfusions - who are clinically stable for at least 1 month before study entry.

Exclusion Criteria: - Patients having a history of any important blood disease - having any clinically significant disease or malfunction of the lungs, heart, hormones, neurological, gastrointestinal, reproductive or urinary systems, which is not caused by the AIDS infection - having dementia due to AIDS, a history of seizures, uncontrolled high blood pressure, or an iron deficiency - androgen therapy within 2 months of study entry - having anemia caused by other conditions than AIDS or AZT therapy (for example, certain vitamin deficiencies or bleeding from the gastrointestinal tract) - having a sudden onset of infections, or a history of cell damage due to chemotherapy within 1 month before study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 1988-07; Study Completion 1990-04 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin and hematocrit (laboratory tests used to evaluate the severity of anemia); Transfusion requirements; Patient's quality of life assessment

SECONDARY OUTCOMES:
Adverse events; changes in clinical laboratory tests, vital signs, electrocardiograms, and physical examination findings; Physician's global evaluation of the overall effect of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech, Inc.

REFERENCES:
- See also: A Study to Evaluate the Safety and Efficacy of Epoetin Alfa in Patients with Acquired Immune Deficiency Syndrome (AIDS) Who Are Receiving AZT Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=709&filename=CR006076_CSR.pdf
- See also: A Study to Evaluate the Safety and Efficacy of Epoetin Alfa in Patients with Acquired Immune Deficiency Syndrome (AIDS) Who Are Receiving AZT Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=709&filename=CR006076_CSR1.pdf